CLINICAL TRIAL: NCT00001610
Title: Normal Human Electro-Oculogram
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970080; 97-EI-0080
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-03

CONDITIONS: Healthy
Keywords: Standing Potential; Fast Oscillation; Slow Oscillation; Retinal Pigment; Epithelium; Electro-oculogram; Cellular Immune Response; Retinal Antigens; IRBP; S-Antigen; Normal Volunteer

SUMMARY:
This study will measure the normal range of the human electro-oculogram (EOG) in people of various age groups. EOGs are recordings of electrical signals generated by the retina (the light-sensitive tissue in the back of the eye) when going from a dark to a bright environment. They provide valuable information about the function of the eye in health and disease. A knowledge of what results are to be expected in tests of normal, healthy eyes will be valuable in assessing EOG results in patients with known or suspected retinal diseases.

Normal volunteers from ages 6 to 65 who have healthy eyes and normal eyesight will participate in this study. Candidates will undergo tests to check vision and the health of the eye. Study participants will then have an electro-oculogram. In this test, eye drops are placed in the eye to enlarge the pupils. Two electrodes (small disks that picks up electrical signals) are attached to the left and right of each eye and one to the forehead. (These are similar to electrodes placed on the body during an electrocardiogram (ECG), which measures electrical signals from the heart.) During the EOG recording, the volunteer looks at the inside of a hollow sphere, following with their eyes small red lights that turn on and off. The background light is also turned on or off during the test. Some volunteers may be asked to repeat the EOG at another time.

Study participants may also be asked to provide a blood sample for tests to study how the immune cells in the blood respond to proteins found in the retina. The response from normal volunteers will be compared with that of patients with eye diseases like retinitis pigmentosa.

DETAILED DESCRIPTION:
Electro-oculograms (EOGs) will be recorded in volunteers of different age groups with normal visual function. The fast and slow oscillations of the EOG will be studied. For the analysis of fast EOG oscillations, peak-to-peak amplitude (micro V), peak-to-trough ratio, and phase (degrees) will be measured. The analysis of slow EOG oscillations will include measurements of the ratio of light peak to dark trough (Arden ratio), implicit time (latency) of the light peak (ms), and amplitude of the dark trough (micro V).

ELIGIBILITY:
Subjects must have best corrected visual acuity equal or better than 20/20.

Subjects must have normal visual fields.

Subjects must have normal color vision.

Subjects must have a normal ophthalmological exam.

Subjects should not be subjective to or objective evidence of visual loss.

Subjects cannot have subjective evidence of abnormal night vision or subjective evidence of abnormal light sensitivity.

Subjects cannot have a personal history of non-trivial ocular disease.

Subjects cannot have a family history of hereditary ocular disease.

Subjects cannot have current systemic disease.

Subjects cannot currently take neuropharmacological medication.

Subjects will not be admitted with an abnormal ophthalmological examination.

Subjects will need the ability to cooperate with EOG recording.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1997-02; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Guideline nine: guidelines on evoked potentials. American Electroencephalographic Society. J Clin Neurophysiol. 1994 Jan;11(1):40-73. No abstract available. PMID 8195426
- [Background] Steinberg RH. Interactions between the retinal pigment epithelium and the neural retina. Doc Ophthalmol. 1985 Oct 15;60(4):327-46. doi: 10.1007/BF00158922. PMID 3905312
- [Background] Marmor MF, Zrenner E. Standard for clinical electro-oculography. International Society for Clinical Electrophysiology of Vision. Arch Ophthalmol. 1993 May;111(5):601-4. doi: 10.1001/archopht.1993.01090050035023. PMID 8489436